CLINICAL TRIAL: NCT02032368
Title: Decrease in Circulating Tumour Cell Count Reflects the Effectiveness of Postoperative Adjuvant Transarterial Chemoembolization (TACE) in Preventing Hepatocellular Carcinoma Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CTCtrial001
Record Dates: First submitted 2014-01-06; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Circulating Tumor Cell;; Hepatocellular Carcinoma
Keywords: circulating tumour cell;; transarterial chemoembolization;; hepatocellular carcinoma;; recurrence
MeSH Terms: conditions — Neoplastic Cells, Circulating; Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE group (Experimental): Patients in TACE group receive transarterial chemoembolization (TACE) one month after resection.
  Interventions: Procedure: transarterial chemoembolization (TACE)
- Control group (No Intervention): Patients in Control group receive no management.

INTERVENTIONS:
Procedure: transarterial chemoembolization (TACE)
  Arms: TACE group

SUMMARY:
Circulating tumour cell (CTC) count could reflect the effect of postoperative transarterial chemoembolization (TACE) on hepatocellular carcinoma (HCC) recurrence.

DETAILED DESCRIPTION:
Early metastases of hepatocellular carcinoma (HCC) may be detected by the isolation of circulating tumor cells (CTCs) in the bloodstream. During the course of therapeutic attempts, monitoring CTC changes in patients with HCC is helpful for the efficacy assessment. Nevertheless, the markers used for the detection, such as a-feto protein, asialoglycoprotein receptor or epithelial cell adhesion molecule, CD133 or CD90, are not specific for HCC CTCs. In spite of these limitations, a timely determination of the existence of CTCs will be beneficial for the monitoring of distant metastases, the evaluation of therapeutic attempts, and the prediction of prognosis.

ELIGIBILITY:
Inclusion Criteria:

* definitive pathological diagnosis of HCC based on World Health Organization (WHO) criteria;
* underwent curative resection one month ago, CT or MRI detecting no new lesions when recruited;
* CTC counts≥2 after resection;
* age between 18 and 75 years;
* adequate hematologic function (platelet count: >60 × 109 platelets/L; hemoglobin: >90g/L; and prothrombin time: <3 seconds above control);
* adequate renal function (serum creatinine: ≤1.5 × upper limit of normal);
* Child-Pugh classification A or B grade

Exclusion Criteria:

* a hypovascular tumor (defined as a tumor with all its parts less contrast-enhanced than the nontumorous liver parenchyma on arterial phase computed tomography scans);
* diffuse-type HCC;
* evidence of hepatic decompensation including esophageal or gastric variceal bleeding or hepatic encephalopathy;
* severe underlying cardiac or renal diseases;
* color Doppler ultrasonography showing portal vein tumor thrombosis with complete main portal vein obstruction without cavernous transformation;
* obstructive jaundice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change of circulating tumor cell(CTC) count at different timepoints | time before TACE and time after TACE
  The time points for blood collection to count CTC were1)one day before TACE(also one month after resection);2)three days after TACE;3)one month after TACE;4) two months after TACE;5)three months after TACE;6)six months after TACE;7) one year after TACE.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Interventional Radiology; Cancer Center; Guangdong General Hospital, Guangzhou, Guangdong, China